CLINICAL TRIAL: NCT06858722
Title: Safety and Efficacy of Ripertamab in Patients with Chronic Inflammatory Demyelinating Polyneuropathy (RIPERT-CIDP): a Randomised, Double-blind, Multicentre, Placebo-controlled Phase 3 Trial
Brief Title: Ripertamab for the Treatment of Chronic Inflammatory Demyelinating Polyneuropathy
Acronym: RIPERT-CIDP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-347-02
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: ripertamab
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ripertamab — On Day 1 of the treatment period, an intravenous infusion of Ripertamab at a dose of 375 mg/m² body surface area will be administered.
  Arms: Treatment group
Drug: Placebo — On Day 1 of the treatment period, an intravenous infusion of Placebo at a dose of 375 mg/m² body surface area will be administered.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if ripertamab works to treat chronic inflammatory demyelinating polyneuropathy. It will also learn about the safety of ripertamab. The main questions it aims to answer are:

Does ripertamab reduce the risk of recurrence in patients? What medical problems do participants have when taking ripertamab? Researchers will compare ripertamab to a placebo (a look-alike substance that contains no drug) to see if ripertamab works to treat chronic inflammatory demyelinating polyneuropathy.

Participants will:

A single intravenous infusion of drug ABC or placebo. Visit the clinic for checkups and tests during W1, W2, W4, W8, W12 Keep a diary of their symptoms and the number of times they undergo rescue therapy

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the requirements of the trial, provide written informed consent (including consent to use and disclose health information related to the study), and willing and able to comply with the trial protocol procedures (including required trial visits);
2. Aged 18 years or older at the time of signing the informed consent form;
3. Diagnosed with definite CIDP according to the 2021 EFNS/PNS criteria;
4. CIDP Disease Activity Status (CDAS) score of ≥2 at screening;
5. INCAT score of at least 2 at initial screening;
6. Meet one of the following conditions: currently receiving oral corticosteroid therapy (equivalent to prednisone/ prednisolone ≤10 mg/day), and/or intravenous immunoglobulin (IVIg) or subcutaneous immunoglobulin (SCIg), but willing to discontinue this treatment before screening; or untreated: no prior treatment; or discontinued corticosteroids and/or IVIg or SCIg at least 6 months before screening;
7. Women of childbearing potential with a negative pregnancy test at screening and a negative urine pregnancy test at baseline;
8. Women of childbearing potential must use a highly effective contraceptive method (failure rate less than 1% per year) from screening until 90 days after the last administration of the investigational medicinal product (IMP);
9. Men who are not surgically sterile and have partners of childbearing potential must use condoms, and their partners must use a highly effective contraceptive method from screening until 90 days after the last administration of the IMP (failure rate less than 1% per year). Men who are surgically sterile (documented azoospermia following vasectomy) may be included. In addition, men must not donate sperm from screening until 90 days after the last administration of the IMP.

Exclusion Criteria:

1. Pure sensory atypical CIDP (defined by EFNS/PNS criteria);
2. Polyneuropathy due to other causes, including but not limited to: multifocal motor neuropathy, monoclonal gammopathy of undetermined significance caused by anti-myelin-associated glycoprotein immunoglobulin M antibodies, hereditary demyelinating neuropathy, polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes syndrome, lumbosacral radiculoplexus neuropathy, polyneuropathy most likely caused by diabetes, polyneuropathy most likely caused by systemic disease, polyneuropathy caused by drugs or toxins;
3. Any disease that can better explain the patient's symptoms and signs;
4. History of any myelopathy or evidence of central demyelination;
5. Current or past (within 12 months before screening) history of alcohol, drug, or substance abuse;
6. Severe psychiatric disorder (e.g., major depression, psychosis, bipolar disorder), history of suicide attempt, or current suicidal ideation that the investigator believes may pose undue risk to the patient or affect the patient's ability to comply with the trial protocol;
7. Clinically significant active or chronic uncontrolled bacterial, viral, or fungal infections at screening, including patients with active viral infections detected at screening: active hepatitis B virus (serological tests indicate active [acute or chronic] infection), active hepatitis C virus (HCV) (HCV-Ab seropositive), human immunodeficiency virus seropositive with acquired immunodeficiency syndrome-defining conditions or CD4 count ≤200 cells/mm³;
8. Total immunoglobulin G level <6 g/L at screening;
9. Received the following treatments: within 1 month before screening (or five half-lives of the drug, whichever is longer): plasmapheresis or immunoadsorption, or any other investigational product; within 6 months before screening: any anti-CD20 monoclonal antibody or other biologic (e.g., rituximab), alemtuzumab, any other monoclonal antibody, cyclophosphamide, interferon, tumor necrosis factor-α inhibitor, fingolimod, methotrexate, azathioprine, mycophenolate mofetil, any other immunomodulatory or immunosuppressive drug, and oral daily corticosteroids >10 mg/day (patients using IVIg, SCIg, corticosteroid pulse therapy, and oral daily corticosteroids ≤10 mg/day may be included);
10. Pregnant and breastfeeding women, and those who plan to become pregnant during the trial or within 90 days after the last dose;
11. Any other known autoimmune disease that the investigator believes may interfere with the accurate assessment of CIDP clinical symptoms;
12. Received live attenuated vaccines within 28 days before screening (patients who received inactivated, subunit, polysaccharide, or conjugate vaccines at any time before screening are not considered exclusion criteria);
13. History of malignancy, unless the patient has been free of recurrence for ≥3 years after adequate treatment before the first dose. Patients with the following cancers may be included at any time: adequately treated basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast, or prostate cancer (tumor, node, and metastasis stage T1a or T1b);
14. Patients who have previously participated in a Ripertamab trial and received ≥1 dose of Ripertamab;
15. Patients with a history of known hypersensitivity to any component of Ripertamab;
16. Any other significant severe disease, or recent major surgery or planned major surgery, or any other reason that may confound trial results or pose undue risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The time to first increase of ≥1 point in the aINCAT score compared to baseline. | Within 24 weeks